CLINICAL TRIAL: NCT04590170
Title: French Cohort of covid19 Patients With Post-intensive Care Syndrome : Rehabilitation From Intensive Care Unit to Home Return - Spatio-temporal Analysis of Walking Compared to Asymptomatic Participants
Brief Title: French Cohort of COVID-19 Patients With Post-intensive Care Syndrome
Acronym: COREADOM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200812
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Covid19 infection: Patients with Covid19 infection
  Interventions: Behavioral: Post-intensive Care unit syndrome
- Control group: Asymptomatic group
  Interventions: Other: Spatiotemporal measurements of walking

INTERVENTIONS:
Behavioral: Post-intensive Care unit syndrome — Post-intensive Care unit syndrome after an intensive care unit stay for the COVID19
  Groups: Patients with Covid19 infection
Other: Spatiotemporal measurements of walking — Spatiotemporal measurements of walking in asymptomatic participants from the general population.
  Groups: Control group

SUMMARY:
The purpose of this study is to describe post-intensive care syndrome (PICS) of patients surviving to coronavirus disease 2019 (COVID19) and their rehabilitation and recovery process from hospital to home return

DETAILED DESCRIPTION:
The novel coronavirus, Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) causing the COVID-19 emerged in December 2019 and was declared pandemic in March 2020.

Although the majority of reported COVID-19 cases are mild, approximatively 5% of patients require a stay in intensive care unit, with mechanical ventilation.

Post intensive care syndrome (PICS) consists of physical, cognitive and psychological dysfunctions.

Little is known about the rate and clinical presentations of PCIS among patients surviving to COVID-19.

The objective of this study is to describe the clinical manifestations of PCIS in COVID-19 patients, and their rehabilitation process until home return.

ELIGIBILITY:
Inclusion Criteria - patients with covid19 infection :

* COVID 19 infection (PCR or CT-scan)
* ICU stay requiring mechanical ventilation
* Age ≥18 years old

Inclusion Criteria - control group :

* Age ≥ 18 years old
* Able to walk without technical assistance,
* Having no orthopedic or neurological disorder likely to disturb balance and walking
* Have not had a severe form of Covid 19 disease in the last 12 months
* Collection of non-opposition

Exclusion Criteria:

- Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in cochin or Corentin-celton hospitals after an intensive care unit stay for a COVID19 infection
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change on cognitive Impairment: Vigilance (RASS) | Between 10 days and 1 month after ICU's discharge
  Used to measure the agitation or sedation level of a person. Range -5 to +4 - Patients group
Change on cognitive Impairment: Cooperation | Between 10 days and 1 month after ICU's discharge
  Yes/no - Patients group
Change on cognitive Impairment: Communication | Between 10 days and 1 month after ICU's discharge
  Yes/no - Patients group
Change on cognitive Impairment: Agitation | Between 10 days and 1 month after ICU's discharge
  Yes/no - Patients group
Change on cognitive Impairment: Delirium | Between 10 days and 1 month after ICU's discharge
  Yes/no - Patients group
Change on cognitive Impairment : Introduction of neuroleptic | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on cognitive Impairment: temporo-spatial disorientation | Between 10 days and 1 month after ICU's discharge
  Yes/no - Patients group
Change on physical Impairment : dyspnea | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/No - Patients group
Change on physical Impairment: Modified Borg scale dyspnea score. | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Verbal and numerical scale that asks you to rate the difficulty of your breathing Patients are asked to tick the boxes that reflect their dyspnea perception best range 0-10 lesser is better - Patients group
Change on physical Impairment : cough | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/No - Patients group
Change on physical Impairment : respiratory rate | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Number of breaths/per minute. - Patients group
Change on physical Impairment : ventilation mode | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Tracheotomy/ ambient air / OXYGEN THERAPY Other - Patients group
Change on physical Impairment : Peripheral capillary oxygen saturation (SpO2) at rest | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  measured by pulse oximetry, which provides an indirect measurement of arterial oxygenation (SaO2) based on the differential absorption of light by oxygenated and deoxygenated blood during pulsatile blood flow - Patients group
Change on physical Impairment : respiratory rate on activity | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  respiratory rate breathing rate on activity - Patients group
Change on physical Impairment : Peripheral capillary oxygen saturation (SpO2) on activity | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  measured by pulse oximetry, which provides an indirect measurement of arterial oxygenation (SaO2) based on the differential absorption of light by oxygenated and deoxygenated blood during pulsatile blood flow during activity - Patients group
Change on physical Impairment : orthostatic hypotension | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no drop in blood pressure that occurs when moving from a laying down (supine) position to a standing (upright) position. - Patients group
Change on physical Impairment : electrocardiogram at rest | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  electrocardiogram at rest - Patients group
Change on physical impairment : numeric verbal scales of fatigue | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  self-evaluation numeric verbal scales of fatigue - Patients group ranges (0-10) lesser is better
Change on physical Impairment: numeric verbal scales of pain | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  self-evaluation numeric verbal scales of pain ranges (0-10) lesser is better
Change on physical Impairment : stiffness or pain involving joints | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/No small joints (wrists, fingers, toes) and large joints (shoulders, elbows, hips, knees, ankles)
  * Patients group
Change on physical Impairment : stability of the trunk in siting | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on physical Impairment : autonomy for bed-chair transfers | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on physical Impairment autonomy for walking | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on physical Impairment : sores | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no Localisation
  * Patients group
Change on Imagery cerebral | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  date and result if applicable - Patients group
Change on physical Impairment neurologic exam | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  motor or sensory deficits involving the upper and the lower limbs (yes/no) Anosmia Yes/no taste loss Yes/no
  * Patients group
Change on physical Impairment Medical Research Council (MRC-SS MRC Sum score) | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  assess muscle strength from Grade 5 (normal) to Grade 0 (no visible contraction).
  MRC-SS score was defined as the sum of MRC scores from six muscles in the upper and lower limbs on both sides so that the score ranged from 60 (normal) to 0 (quadriplegic).
  * Patients group
Change on physical Impairment five times sit to stand test | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times without use of arms, Equipment • Standard height chair (43-45 cm, 17-18 inches) with a backrest. If the patient cannot perform five stands to complete the test without use of arms, a score of 0 seconds should be documented.
  * Patients group
Change on cognitive Impairment The Montreal Cognitive Assessment (MoCA) | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstruction skills, conceptual thinking, calculations, and orientation. Range 0 -30 higher is better
  * Patients group
Cognitive Impairment Frontal Assessment Battery (FAB) | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Total score is from a maximum of 18, higher scores indicating better performance.
  * Patients group
Change on psychological Impairment : sadness | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : anxiety | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment: Insomnia | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : Apathy | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : sideration | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : Despair | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : Culpability | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : Conduit addictive | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
Change on psychological Impairment : psychiatric or psychologic care | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Yes/no - Patients group
assess type of psychiatric treatment | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Type - Patients group
Change on psychological Impairment : Hospital Anxiety and Depression Scale (HADS) | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  A 14-item self-report screening scale that was originally developed to indicate the possible presence of anxiety and depressive states It contains two 7-item scales: one for anxiety and one for depression both with a score range of 0-21.
  * Patients group
Change on psychological Impairment : Posttraumatic Stress Disorder Checklist Scale (PCL-S) | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  20-item questionnaire, corresponding to the Manual of Mental Disorders (DSM-5) symptom criteria for PTSD.
  * Patients group
assess psychological Impairment | Change between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Introduction of antidepressant drugs Type
  * Patients group
assess psychological Impairment | change between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Introduction of neuroleptic Type
  * Patients group

SECONDARY OUTCOMES:
asses demographics information | Between 10 days and 1 month after ICU's discharge
  Age, sex, formal education, marital status, occupation, place of living, socio-professional category
  * Patients group
assess comorbidities | Between 10 days and 1 month after ICU's discharge
  number of comorbidities
  * Patients group
assess past and current medications | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Precise
  * Patients group
assess related symptoms nature of COVID-19 | Between 10 days and 1 month after ICU's discharge
  duration of COVID-19-related symptoms nature Laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay and/or CT-scan showing typical radiological findings
  * Patients group
assess characteristics of ongoing hospitalization | Between 10 days and 1 month after ICU's discharge
  number of characteristics of ongoing hospitalization (invasive ventilation, curare, others treatments )
  * Patients group
assess medical complications in intensive care | Between 10 days and 1 month after ICU's discharge
  Pneumopathy pulmonary embolism others
  * Patients group
Descriptive data of the rehabilitation care pathway after stay in intensive care until return home | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  Number of days to discharge from hospital Service of rehabilitation care hospital at home (HAH) return at home
  * Patients group
Number of new medical qualifying events since last contact | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  complications
  * Patients group
Social status | Between 10 days and 1 month and 3 months and 6 months after ICU's discharge
  professional activity unemployment retirement others
  * Patients group
Activities of Daily Living (ADL) scale | 3 months and 6 months after ICU's discharge
  Related to personal care (self-performance) looks at four of these tasks: transfer, bed mobility, toileting and eating. The resident's self- performance and the amount of staff support provided are evaluated for all of these tasks ranges from 0 (independent) to 4 (total dependence)
  * Patients group
Quality of life Medical outcome study short form 12 items (MOS-SF-12 ) questionnaire | 3 months and 6 months after ICU's discharge
  Self-reported outcome measure assessing the impact of health on an individual's everyday life Patients fill out a 12-question survey which is then scored by a clinician or researcher.
  Questionnaire consisting of 12 questions that measure 8 health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH).
  * Patients group
Gait analysis 6-minute walk test (6MWT) | 3 months and 6 months after ICU's discharge
  Sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
  * Patients group
Balance and Gait analysis | 3 months and 6 months after ICU's discharge
  Inertial Sensors to Assess Gait Quality
  * Patients group
Spatio-temporal parameters of walking | Inclusion
  Comparison of spatio-temporal measures of walking in patients with severe Covid 19 infection to those of an age- and sex-matched sample of asymptomatic participants.
  Both groups

CONTACTS AND LOCATIONS:
Overall Officials: Camille DASTE, MD, Principal Investigator — Study Principal Investigator
Locations (2):
- France (2):
  - Department of Rehabilitation, Institute of Rheumatology Cochin, Paris, Paris
  - Department of Physical Medicine and Rehabilitation, Issy-les-Moulineaux

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daste C, Ficarra S, Dumitrache A, Cariou A, Lefebvre A, Pene F, Roche N, Roren A, Thery C, Vidal J, Nguyen C, Rannou F, Lefevre-Colau MM. Post-intensive care syndrome in patients surviving COVID-19. Ann Phys Rehabil Med. 2021 Nov;64(6):101549. doi: 10.1016/j.rehab.2021.101549. Epub 2021 Jun 26. No abstract available. PMID 34182168